CLINICAL TRIAL: NCT00053599
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial of Simvastatin to Slow the Progression of Alzheimer's Disease
Brief Title: Cholesterol Lowering Agent to Slow Progression (CLASP) of Alzheimer's Disease Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0038; ADC-015-LL
Record Dates: First submitted 2003-02-03; First posted 2003-02-04 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-06

CONDITIONS: Alzheimer Disease
Keywords: Cholesterol-lowering drug; Mild to Moderate Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
CLASP is a research study to investigate the safety and effectiveness of simvastatin (a cholesterol lowering drug or statin) to slow the progression of Alzheimer's disease (AD). Statins are commonly used to treat high cholesterol levels, which increase the risk of heart disease and stroke.

DETAILED DESCRIPTION:
In earlier studies in animals and humans, researchers found that lowering cholesterol levels with statins seems to have a positive impact on brain function and reduces the risk of AD. The CLASP trial will test the link between using a cholesterol lowering medication and slowing disease progress in people with mild to moderate Alzheimer's disease (AD).

CLASP is a research study to investigate the safety and effectiveness of simvastatin (a cholesterol lowering drug or statin) to slow the progression of AD. The clinical trial will include the treatment of patients with mild to moderate AD, and the objective is to evaluate the safety and efficacy of simvastatin to slow the progression of AD, as measured by the cognitive portion of the AD Assessment Scale. Measures of clinical global change (ADCS-CGIC), mental status, functional ability, behavioral disturbances, quality of life and economic indicators will be made also. The study design is randomized, double-blind, placebo-controlled, parallel group design with equal randomization to drug and placebo. Randomization will be stratified and blocked to ensure balanced assignment within site. Sample size will include 400 participants enrolled from approximately 40 sites with a goal of 10 to 15 volunteers enrolled at each site. Study medication will be as follows: 20 mg of simvastatin or matching placebo to be given for 6 weeks, followed by 40 mg of simvastatin or matching placebo for the remainder of the 18-month study period. Participants will be instructed to take the medication once a day in the evening. Safety parameters to be checked will include adverse events, symptom checklists, vital signs, physical and neurological examinations, and laboratory tests.

ELIGIBILITY:
* Mild to moderate patients with AD who are free of life-threatening disease and who do not require lipid-lowering treatment according to current guidelines.
* NINCDS/ADRDA criteria for probable AD.
* Mini-Mental-State-Exam (MMSE) score between 12 and 26.
* Stable medical condition for 3 months prior to the screening visit.
* Age greater than or equal to 50 years, and no upper age limit.
* Lives in a community dwelling, not in a nursing home.
* Stable doses of (non-excluded) medications with central nervous system activity for 4 weeks prior to the screening visit.
* Physical condition acceptable for the study as confirmed by medical history, physical exam, neurologic exam and clinical laboratory tests.
* Informant/study partner available and willing to accompany participant to all scheduled visits and complete informant-based assessments and to supervise administration of study medications.
* Fluent in English or Spanish.
* Modified Hachinski is less than or equal to 4.

Exclusion criteria:

* Coronary heart disease (CHD) including angina, or peripheral vascular disease including symptomatic carotid artery disease, or stroke or TIA, as these individuals are likely to require treatment with lipid-lowering drugs.
* Serious renal disease.
* Uncontrolled diabetes.
* Triglycerides are greater than 500 mg/dL.
* LDL-Cholesterol below 80 mg/dL
* Upper limit for the National Cholesterol Education Program (NCEP) guidelines for LDL-Cholesterol is 130-190 mg/dL, depending on age and other cardiovascular risk factors.
* Other indication for the need to treat with lipid-lowering drug.
* Active liver disease or persistent elevation in serum transaminase.
* Active neoplastic disease (skin tumors other than melanoma are not exclusionary; subjects with stable prostate cancer may be included at the discretion of the Project Director).
* Use of another investigational agent within 2 months of the screening visit.
* History of clinically significant stroke.
* Current evidence or history in the past 2 years of seizures, head injury with loss of consciousness and/or immediate confusion after the injury.
* Current DSM-IV criteria based diagnosis for major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse.
* Blindness, deafness, language difficulties or any other disability which may prevent the subject from participating or cooperating in the protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2002-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sano, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Leon J. Thal, MD, Principal Investigator — University of California, San Diego
Locations (44):
- United States (44):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Barrow Neurology Group, Phoenix, Arizona
  - Arizona Health Sciences Center, University of Arizona, Tucson, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University/VA Aging Clinical Research Center, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Memory Disorder Program, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Baumel Eisner Neuromedical Institute, Boca Raton, Florida
  - Mayo Clinic (Jacksonville), Jacksonville, Florida
  - Wein Center, Miami Beach, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush Alzheimer's Disease Center, Rush University, Chicago, Illinois
  - Indiana University Alzheimer's Center, Indianapolis, Indiana
  - University of Kentucky, Sanders-Brown Center on Aging, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan at Ann Arbor, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - Washington University, St. Louis School of Medicine, St Louis, Missouri
  - SUNY Downstate, Brooklyn, New York
  - New York University School Of Medicine, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Neurological Care of NY, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Memory and Aging Center, Case Western Reserve University/University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania School of Medicine, Alzheimer's Disease Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University-Memorial Hospital of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - University of Texas, Southwestern Medical School, Dallas, Texas
  - Baylor College of Medicine, Alzheimer's Disease Research Center, Houston, Texas
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - University of Washington at Seattle, Seattle, Washington

REFERENCES:
- [Background] Hartmann T. Cholesterol, A beta and Alzheimer's disease. Trends Neurosci. 2001 Nov;24(11 Suppl):S45-8. doi: 10.1016/s0166-2236(00)01990-1. PMID 11881745
- [Background] Jick H, Zornberg GL, Jick SS, Seshadri S, Drachman DA. Statins and the risk of dementia. Lancet. 2000 Nov 11;356(9242):1627-31. doi: 10.1016/s0140-6736(00)03155-x. PMID 11089820
- [Background] Simons M, Schwarzler F, Lutjohann D, von Bergmann K, Beyreuther K, Dichgans J, Wormstall H, Hartmann T, Schulz JB. Treatment with simvastatin in normocholesterolemic patients with Alzheimer's disease: A 26-week randomized, placebo-controlled, double-blind trial. Ann Neurol. 2002 Sep;52(3):346-50. doi: 10.1002/ana.10292. PMID 12205648
- See also: Alzheimer's Disease Cooperative Study — http://www.adcs.org/